CLINICAL TRIAL: NCT06019806
Title: Effects of Forward Head Posture Correction on Visual Acuity and Fatigue in Low Level Visually Impaired University Students
Brief Title: Effects of Forward Head Posture Correction on Visual Acuity in Low Level Visually Impaired University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RiphahIU Shabi ul Hassan
Record Dates: First submitted 2023-08-26; First posted 2023-08-31 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Visual Acuity
Keywords: forward head posture; visual fatigue; craniovertebral angle; postural correction exercises
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postural correction group A (Experimental): 1. Chin tuck (deep cervical flexor)
  2. Strengthening shoulder retractors
  3. Sternocleidomastoid muscle stretch
  4. Pectoralis stretch
  Interventions: Other: POSTURAL CORRECTION four exercises
- Control group B (Active Comparator): postural Correction education
  Interventions: Other: postural Correction education with a manuscript

INTERVENTIONS:
Other: POSTURAL CORRECTION four exercises — The program will involve four exercises, including two strengthening exercises and two stretching exercises.
  1. Chin tuck (deep cervical flexor)
  2. Strengthening shoulder retractors
  3. Sternocleidomastoid muscle stretch
  4. Pectoralis stretch Participants will be instructed to perform three sets of 12 repetitions for the strengthening exercises, with a 30-second rest period allotted between each set. For the stretching exercises, participants will be instructed to hold each stretch for 30 seconds, with a 30-second rest period allotted between each exercise The experimental group will also receive postural Correction education
  Arms: postural correction group A
Other: postural Correction education with a manuscript — The control group would receive postural Correction education and they would be provided with a manuscript. They would be then guided to follow these guidelines as a home plan for four weeks. At the end of the Fourth week, they would be assessed.
  Arms: Control group B

SUMMARY:
The aim of this research is to find the effect of forward head posture correction on visual acuity and fatigue in low level visually impaired university students. Randomized controlled trials at Cecos University of IT and Emerging Sciences would be done. The sample size would be 48. The subjects would be divided in two groups, 24 subjects Intervention group and 24 in control group. Study duration would be 6 months. Sampling technique applied would be a non-probability convenience sampling technique. Only 18-25 years low level visually impaired university students with forward head posture would be included. Tools used in the study would be asthenopia questionnaire, Snellen chart and CVA angle photogrammetry

DETAILED DESCRIPTION:
In recent years, the increasing use of modern technology has raised concerns about its potential impact on our visual health. However, research suggests that in addition to these factors environmental factors such as near work, visual stress, educational stress and acquired false head posture may have a greater impact on visual health of young adult population. Prolonged use of digital devices can cause digital eye strain, leading to symptoms such as headaches and blurred vision. However, poor posture can also cause strain on the eyes, leading to decreased visual acuity and compromised performance. It is essential to consider factors such as posture when assessing visual performance in university students, in addition to the impact of modern technology. The forward head posture (FHP) is the head movement that occurs from poor postural awareness and frequently leads to muscle imbalance and discomfort.

University students frequently experience a forward head position, especially those who spend a lot of time studying or using computers. Both forward head posture and visual impairment are more prevalent among university students. It has been found that 63.96% of university students, including both genders, exhibit a prevalence of forward head posture. . A 2019 study in America found that 67.8% of university students experience visual fatigue, with blurred vision being the most commonly reported symptom (27%). This suggests many students may have mild visual impairments, impacting their academic performance and quality of life. The existing research has mainly concentrated on studying visual impairment by defining specific levels of impairment such as 'moderate' and 'severe.' However, it is plausible that even a minor reduction in visual acuity, also known as 'mild' visual impairment (ranging from 20/30 to 20/70), could have a subtle but significant impact on an individual's ability to cope with activities of daily life. The position and movement of the head play a crucial role in visual perception, as the somatosensory system of the neck is intricately connected to the visual system. Spending most of the time using computers, mobile phones and reading can cause biomechanical alterations that make it difficult to keep a neutral head position and compromise the structural integrity .The Centre of Gravity (COG) of the head moves in anterosuperior direction as a result of this structural integrity compromise, increasing the stress on the neck. Each inch that the head is moved forward or anteriorly from its neutral position adds approximately 10 pounds (4.5 kilograms) of extra weight to the cervical spine.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Mild visual impairment, visual acuity of 20/30 to 20/70 and with symptoms of visual fatigue
* Forward head posture (FHP)
* Craniovertebral Angle less than 48-50
* Able to understand and provide informed consent
* Able to participate in the intervention and attend all the required

Exclusion Criteria:

* Visual impairment other than mild visual impairment (e.g., legal blindness)
* Pre-existing medical conditions or injuries that may affect the posture or visual function
* Any previous neck and Eye surgery.
* Previous history of treatment for FHP or visual impairment in the past six months(23)
* Any physical, neurological or cognitive disability that may affect the ability to participate in the intervention or the assessments
* Use of medication or treatments that may affect the posture or visual function
* Psychological conditions

Ages: 15 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Snellen Chart | 4 weeks
  Universally used for measuring visual acuity.
Asthenopia Questionnaire | 4 weeks
  Used for measuring Visual fatigue.
Craniovertebral Angle | 4 weeks
  Craniovertebral angle is measured by taking 2 lateral photographs of the subject in a relaxed seated position without a back support. Spinous process of C7 and the tragus of ear are marked with a body marker. A horizontal line is drawn passing through C7 making a right angle with the vertical.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Cecos University of IT and Emerging Scienecs, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No